CLINICAL TRIAL: NCT06402383
Title: Supporting the National Expansion of HPV-based Cervical Cancer Screening in Tanzania Among Women Living with HIV: NECST-HIV
Brief Title: Supporting the National Expansion of HPV-based Cervical Cancer Screening in Tanzania Among Women Living with HIV
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Merck Canada Inc. (Industry)
Responsible Party: Principal Investigator, Dr. Karen Yeates, Professor, Queen's University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 102030
Record Dates: First submitted 2024-04-05; First posted 2024-05-07 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Cervical Cancer
Keywords: cervical cancer; cancer prevention; screening
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vaccination starting from visit 1 (Experimental): Vaccination will be provided at the first visit and then at 6 months for HPV negative women and 12 months for HPV positive women.
  Interventions: Biological: Vaccination Provision
- Vaccination starting at follow up (Experimental): Vaccination will be provided after HPV results obtained - immediately for HPV negative women and again after 3 months. For HPV positive women this will be offered at 12 months after testing and again at 15 months.
  Interventions: Biological: Vaccination Provision 2

INTERVENTIONS:
Biological: Vaccination Provision — HPV vaccination #1 will be offered by provider at the first visit when the HPV self-sample is collected. HPV Vaccination #2 will be offered at 6 months for HPV negative women and at 12 months for HPV positive women.
  Arms: Vaccination starting from visit 1
Biological: Vaccination Provision 2 — HPV vaccination #1 will be offered by the provider after an HPV negative result is received with vaccine #2 given at 3 months after negative test results obtained.
  For HPV positive women - vaccination #1 will be offered at 12 months and vaccination #2 will be offered at the 15 month mark.
  Arms: Vaccination starting at follow up

SUMMARY:
* Cervical cancer is caused by persistent infections with one of ~13 carcinogenic human papillomavirus (HPV) types and causes substantial morbidity and mortality worldwide.
* Highly effective strategies exist, including HPV vaccination and HPV-based screening for early detection and treatment of precancerous lesions.
* The investigators are proposing an innovative implementation research program and randomized trial evaluating HPV DNA testing as a primary screening tool for cervical cancer screening in HIV Care and Treatment clinics within Tanzania's National Cervical Cancer Prevention (CECAP) program.
* The investigators will combine HPV DNA testing with high quality visual assessment of the cervix for treatment and management of cervical precancerous lesions among HPV+ Women Living with HIV (WLWH).
* At 12-month follow up women will be recalled for repeat screening for HPV and visual assessment of the cervix for treatment combined with a second therapeutic dose of HPV vaccine.
* The investigators propose to recruit 2000 WLWH from 4 HIV Clinics in Kilimanjaro Region. Two clinics will be randomized to the test, treat and vaccinate strategy and two clinics will be randomized to test, treat and re-screen and then vaccinate strategy.
* Currently, there is no Standard of Care (SOC) for vaccination of women who are at risk for HPV in the country. These two arms of the study will allow for treatment and observation to occur that would not be available otherwise.

ELIGIBILITY:
Inclusion Criteria:

* Gender: person with an intact cervix
* HIV type 1 (HIV-1) positive status and receiving care at one of the study CTC sites randomized for the trial
* Not pregnant and utilizing contraception if sexually active and willing to undergo a urine pregnancy test prior to enrolment
* Residence in the study-defined catchment area
* Willing to consent to receive follow-up phone calls from the health provider to provide reminders and counselling about follow-up visits required for the study procedures
* Willing to receive HPV Vaccination in a 2-dose strategy
* Language: able to speak/understand English or Kiswahili (if the participant cannot read, the consent will be read to her, and thumbprint will suffice for consent as per the Tanzanian National Institute for Medical Research Ethical Guidelines for Informed Consent Processes)

Exclusion Criteria:

* Women will be excluded for a prior history of invasive or microinvasive cervical, vaginal, vulvar, or anal cancer; prior hysterectomy; cervical treatments within 1 year prior to study; cervical, vaginal, or vulvar lesions suspicious for cancer; prior HPV vaccination; receipt of anticoagulants; known sensitivity to vaccine components; hemophilia or bleeding diathesis; use of antineoplastic or immunomodulatory treatment; breastfeeding; and <3 months postpartum. Any potential participant who appears unable to provide informed consent or does not want to participate in the research study will be excluded.

Women that do not want to receive the vaccine will be excluded.

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2000 (Estimated)
Dates: Start 2024-05-25 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Evidence Generation for use of a 4-step HPV testing, triage and vaccinate strategy | 15 months
  The primary endpoint will be a composite of HSIL on cervical histology at 12 months re-screening (follow-up). Secondary endpoints will include CIN3 on cervical histology, and grade 3 or 4 adverse events related to vaccination. Additional secondary endpoints will include participant-level predictors that may act as moderators of participation in cervical cancer screening and/or HPV vaccination. The investigators will also collect qualitative and quantitative data on the feasibility, impact, and cost-effectiveness of the different screening strategies through key informant interviews and focus groups comprised on clinic leadership, health providers and study participants.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Yeates, MD,MPH, Principal Investigator — Queen's University
Locations (1):
- Pamoja Tunaweza Women's Centre, Moshi, Tanzania